CLINICAL TRIAL: NCT04296201
Title: Evaluation of the Immediate Effect and Safety of DMA™ Novel Muscle Stimulation Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUM-ABU-DMA-20-01
Record Dates: First submitted 2020-03-02; First posted 2020-03-05 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Skin Laxity; Muscle Contracture
MeSH Terms: conditions — Cutis Laxa; Contracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Treatment in the face area (Experimental): 5 female subjects will receive treatment in the face area
  Interventions: Device: DMA treatment
- Treatment in the buttocks area (Experimental): 5 female subjects will receive treatment in the buttocks area
  Interventions: Device: DMA treatment
- Treatment in the abdominal region (Experimental): 5 male subjects will receive treatment in the abdominal region
  Interventions: Device: DMA treatment

INTERVENTIONS:
Device: DMA treatment — Each arm will receive the DMA treatment in a specific area on the body to observe immediate effect.

SUMMARY:
A total of at least 15 and up to 17 healthy subjects at a single site, aged 25-45 years old, who wish to receive a lifting effect and improved muscle definition, will be included in the study.

The procedure will include treatments with the Legend Pro™ DMA™ technology. Photos will be obtained at pre-defined time points throughout the study.

DETAILED DESCRIPTION:
Single center, prospective, open Label with Before & After Study Design. This study is designed to evaluate the immediate efficacy and safety of Legend Pro™'s DMA™ muscle stimulation technology. Treatment areas will include the face, buttocks, or abdominal region. Each subject will receive 1 treatment with no follow-up visits required. Interim assessment will be held after half of the study population has received treatment.

The study population will be divided into three arms as follows:

* 5 female subjects will receive treatment in the face area
* 5 female subjects will receive treatment in the buttocks area
* 5 male subjects will receive treatment in the abdominal region

ELIGIBILITY:
Inclusion Criteria:

1. Subject read, understood and signed the Consent Form
2. Healthy male or female aged 25-45 years,
3. Fitzpatrick skin type 1-6
4. Subject is capable of reading, understanding and following instructions of the procedure to be applied.
5. Subject is able and willing to comply with the treatment.
6. Women of child-bearing potential are required to use two forms of reliable methods of birth control (such as an intrauterine device, birth control pills, condom with spermicidal, NuvaRing, partner with vasectomy, Implanon or other FDA-approved devices, or abstinence) during the course of the study.

Exclusion Criteria:

General

1. Subject is female who is pregnant, lactating, or plans to become pregnant during the study period or had given birth less than 6 months ago.
2. Concurrent participation in any other study.

   Specific to the treatment and treatment area
3. Subject has a pacemaker or internal defibrillator, implanted neurostimulators or any other internal electric device or patient who had an implant in the past.
4. Subject has metal or other implants in the treatment area (Not including dental fillings, implants and crowns).
5. Subject has significant concurrent skin conditions affecting areas to be treated such as sores, bleeding, skin fragility, eczema or psoriasis.
6. Subject has burned, blistered, irritated, or sensitive skin due to excessive fresh tanning in areas to be treated or is unlikely to refrain from excessive tanning during the study.

   Other treatments
7. Subject has used oral isotretinoin (Accutane or Roaccutan®) within 6 months prior to study enrollment or plans use during the course of the study.
8. Subject has used topical retinoids in past 1 month

   Medical conditions/ use of medication
9. Subject has current or history of systemic cancer; premalignant skin lesion or skin concern treatment area.
10. Subject has severe concurrent conditions such as epilepsy, autoimmune, pulmonary or cardiac disorders.
11. Subject has poorly controlled endocrine disorders such as diabetes.
12. Subject has an impaired immune system due to immunosuppressive diseases such as HIV or AIDS, or use of immunosuppressive medications.
13. Subject has history of collagen disorders, keloid formation or abnormal wound healing.
14. Subject takes or has taken medications, herbal preparations, food supplements or vitamins that might cause fragile skin or impaired skin healing
15. Subject has used oral steroids in past 6 months
16. Subject has used topical steroids in past 3 months
17. Subject has history of bleeding coagulopathies or use of anticoagulants.
18. Use of non-steroidal anti-inflammatory drugs (NSAIDS, e.g. ibuprofen containing agents) one week before and after each treatment session prior to treatment
19. Subject has mental disorders that in the opinion of the Investigator would be interfere with ability to comply with the study requirements.
20. Subject has any other medical condition that in the opinion of the Investigator warrants exclusion from this study

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
To evaluate the immediate effects and safety of DMATM novel muscle stimulation technology on the face, buttocks, and abdominal regions: GAI scale | 6 months
  Efficacy of the treatment will be based on before and after photography. Efficacy will be established by the Global Aesthetic Improvement scale (GAI) completed by the Principal investigator. Success is defined as an improvement of at least 1 point on the GAI scale assessed by the investigator, as compared to baseline.
  Global Aesthetic Improvement (GAI) Scale:
  Worse (0), No change (1), Somewhat improved (2), Moderately improved (3), Very Much Improved (4)

SECONDARY OUTCOMES:
To evaluate procedure-related skin safety, subject discomfort, and subject satisfaction: questionnaire | 6 months
  The secondary endpoint will be assessed by the following:
  • Subject satisfaction questionnaire
  Safety End-Points:
  * Immediate skin response (erythema, edema, etc.) following each treatment as evaluated by the investigator.
  * Subject assessment of pain and discomfort associated with treatments using a Pain Visual Analogue Scale (VAS), were 0 is "no pain" and 10 is "intolerable pain"
  * Skin safety throughout the study as determined by the investigator by examining the post-treatment occurrences of complications and adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology, Laser, and Vein Specialists of the Carolinas, PLLC, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No